CLINICAL TRIAL: NCT07050043
Title: A Phase III RCT Comparing Low Dose Immunotherapy (Nivolumab) Combined With Standard Chemotherapy vs Standard Chemotherapy as First-line Treatment in Patients With Locally Advanced or Metastatic NSCLC
Brief Title: Low Dose Nivolumab With Chemotherapy vs Standard Chemotherapy as First-Line Treatment in Advanced or Metastatic NSCLC
Acronym: LEDANG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Arvindran A/L Alaga (Other Government)
Responsible Party: Sponsor-Investigator, Dr Arvindran A/L Alaga, Consultant Respiratory Physician, Hospital Sultanah Bahiyah
Organization: Hospital Sultanah Bahiyah (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIT-LEDANG2023001; NIH/800-3/2/2 Jilid 18 (38) (Other Grant/Funding Number: Ministry of Health, Malaysia (MOH))
Record Dates: First submitted 2025-05-15; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: NSCLC (Non-small Cell Lung Carcinoma); First Line Therapy; Locally Advanced/Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Cisplatin; Carboplatin; Pemetrexed; Gemcitabine; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab + Standard Chemotherapy (Experimental): Patient will be receiving of low dose Nivolumab (40mg) combined with standard chemotherapy
  Interventions: Drug: Nivolumab 40mg; Drug: Cisplatin, Carboplatin, Pemetrexed, Gemcitabine, Paclitaxel, Docetaxel
- Standard Chemotherapy (Active Comparator): Patient will be receiving standard chemotherapy alone.
  Interventions: Drug: Cisplatin, Carboplatin, Pemetrexed, Gemcitabine, Paclitaxel, Docetaxel

INTERVENTIONS:
Drug: Nivolumab 40mg — Nivolumab is an immunotherapy medicine used to treat several cancers, including lung cancer.
  Other Names: Opdivo
  Arms: Nivolumab + Standard Chemotherapy
Drug: Cisplatin, Carboplatin, Pemetrexed, Gemcitabine, Paclitaxel, Docetaxel — Cisplatin, carboplatin, pemetrexed, paclitaxel, Gemcitabine, and docetaxel are chemotherapy drugs used to treat various types of cancer, including non-small cell lung cancer.
  Other Names: CDDP; Paraplatin; Taxotere; CBDCA; dFdC; PTX

SUMMARY:
This is a multicenter, two-arm randomized, parallel group design trial to evaluate superiority and safety of low dose Nivolumab (40mg) combined with standard chemotherapy versus standard chemotherapy alone in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Eligible subjects who satisfy the inclusion and exclusion criteria will be randomized 2:1 into 2 arms (Low dose nivolumab arm consisting of six-weekly 40mg Nivolumab plus 4-6* cycles of Cisplatin or Carboplatin plus Pemetrexed or Gemcitabine or Docetaxel or Paclitaxel per local practice, versus standard chemotherapy alone, consisting 4-6* cycles of Cisplatin or Carboplatin plus Pemetrexed or Gemcitabine or Docetaxel or Paclitaxel per local practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent.
2. Histologically confirmed, treatment naïve, locally advanced, or metastatic (stage IIIB - IV (per AJCC version 8), squamous or non-squamous NSCLC with documented PD-L1 expression and is not eligible for definitive chemo-radiation curative therapy and surgery.
3. Patients must be treatment naïve with respect to locally advanced or metastatic disease. Patients who received prior treatment with curative intent for early stage disease and develop recurrent advanced/ metastatic disease must have completed treatment at least 6 months prior to first dose of IP.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
5. At least 1 measurable lesion by RECIST 1.1 in solid tumors criteria.
6. Participants must have adequate organ function including the following laboratory values at the screening visit as per Table 2:
7. If a participant has brain or meningeal metastases, the participant must meet the following criteria:

   1. Metastatic brain lesions do not require immediate intervention. Note: Asymptomatic, treated and stable as well as not requiring steroids for at least 2 weeks prior to start study Treatment.
   2. Carcinomatous meningitis is excluded regardless of clinical stability.
8. A male participant must agree to use a contraception starting with the first dose of study treatment through the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.
9. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP), OR,
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 180 days after the last dose of study treatment.
10. Can provide evaluable archival tumor tissue sample or willing to provide tissue from newly obtained core or excisional biopsy or fine needle aspirate (FNA) cell block form of tumor lesion not previously irradiated. Note: Formalin fixed, paraffin embedded (FFPE) tissue blocks or slides allowed.

Exclusion Criteria:

1. Presence of EGFR, ALK , ROS1 mutation(s).
2. Patients with locally advanced disease who can receive other potentially curative therapies, such as patients who can afford to pay for or can otherwise access clinically approved doses of immunotherapy.
3. Prior treatment with any anti-PD-1, anti-PD-L1 or any other antibody targeting an immune checkpoint.
4. Use of any live vaccines against infectious diseases within 28 days of first dose of IP(s).
5. Underlying medical conditions that, in the Investigator's or Sponsor PI's opinion, will make the administration of IP(s) hazardous, including but not limited to interstitial lung disease, including history of interstitial lung disease or non-infectious pneumonitis (lymphangitic spread of NSCLC is not disqualifying), or active viral, bacterial, or fungal infections requiring parenteral treatment within 14 days of the initiation of the IP.
6. Concurrent medical condition requiring the use of supra-physiologic doses of corticosteroids (> 10 mg/day of oral prednisone or equivalent) or immunosuppressive medications (absorbable topical corticosteroids are not excluded).
7. Active hepatitis B and C infection or human immunodeficiency virus antibody (HIV-1 and/or HIV-2) positive at screening.
8. Known hypersensitivity to recombinant proteins, or any excipient contained in the IP formulations.
9. Known history of autoimmune disease currently on immunosuppressive medications.
10. Known history of second malignancy within two years prior enrolment.
11. Prognosis of three months or less.
12. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment allocation. If the urine test positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From randomization to either the date of progression or death from any cause (whichever comes first) - up to 36 months
  Determine the PFS of six-weekly Nivolumab 40mg combined with standard chemotherapy versus standard chemotherapy alone in NSCLC

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of treatment commencement to the date death from any cause or the date of the last follow-up before final analysis (whichever comes first) - up to 36 months
  Evaluate the OS of six-weekly Nivolumab 40mg combined with standard chemotherapy in NSCLC
Patient-Reported Outcome Measure (PROM) | From the baseline until the end of treatment follow up or the last study follow up related to adverse event - up to 24 months
  Evaluate PROM for six-weekly Nivolumab 40mg combined with standard chemotherapy in NSCLC. For each tool, domain scores and individual scores will be calculated using the scoring or developer's guidelines
PROM using EORTC QLQ-C30 | From the baseline until the end of treatment follow up or the last study follow up related to adverse event - up to 24 months
  A 30-question survey that looks at overall quality of life in cancer patients. It measures five functional dimensions (physical, role, emotional, cognitive, and social), three symptom items (fatigue, nausea/vomiting, and pain), six single items (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact) and global health and quality of life
PROM using EQ-5D-5L | From the baseline until the end of treatment follow up or the last study follow up related to adverse event - up to 24 months
  A 6-question tool to assess general health and well-being through 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
PROM using NSCLC-SAQ | From the baseline until the end of treatment follow up or the last study follow up related to adverse event - up to 24 months
  A 7-question survey that focuses on lung cancer symptoms, including cough, dyspnea, pain, fatigue, and appetite
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose to last dose of treatment plus follow-up - up to 27 months
  To assess the safety and tolerability profile of study regimens, measured by the number and percentage of participants experiencing at least one TEAE, as defined by CTCAE v5.0
Incidence of Serious Adverse Events (SAEs) | From first dose to last dose of treatment plus follow-up - up to 27 months
  To assess the safety and tolerability profile of study regimens, measured by the number and percentage of participants experiencing at least one SAE, as defined by CTCAE v5.0
Incidence of Treatment-Related Discontinuations | From first dose to last dose of treatment plus follow-up - up to 27 months
  To assess the safety and tolerability profile of study regimens, measured by the number and percentage of participants who discontinue treatment due to adverse events, as defined by CTCAE v5.0
Incidence of Treatment-Related Deaths | From first dose to last dose of treatment plus follow-up - up to 27 months
  To assess the safety and tolerability profile of study regimens, measured by the number and percentage of participants who die due to adverse events, as defined by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Arvindran A/L Alaga, Principal Investigator — Hospital Sultanah Bahiyah
Locations (1):
- Hospital Sultanah Bahiyah, Alor Star, Kedah, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT07050043/Prot_000.pdf